CLINICAL TRIAL: NCT02140060
Title: A 6-Week Proof-of-Concept Study Evaluating the Safety and IOP-Lowering Efficacy of Travoprost/Brinzolamide Fixed Combination Ophthalmic Suspension in Subjects With Open-Angle Glaucoma or Ocular Hypertension
Brief Title: 6-Week Proof-of-Concept Study of Travoprost/Brinzolamide Ophthalmic Suspension in Subjects With Open-Angle Glaucoma or Ocular Hypertension
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: C-14-003
Record Dates: First submitted 2014-05-14; First posted 2014-05-16 (Estimated); Results first posted 2015-12-29 (Estimated); Last update posted 2015-12-29 (Estimated); Status verified 2015-11

CONDITIONS: Glaucoma; Ocular Hypertension
Keywords: Glaucoma; Ocular; Hypertension; OAG; POAG; OHT
MeSH Terms: conditions — Glaucoma; Ocular Hypertension; Hypertension | interventions — brinzolamide; Travoprost

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- TravA/Brinz (Experimental): Dose Level A / Brinzolamide 1% ophthalmic suspension (fixed combination), 1 drop twice daily in the treated eye(s) morning and night, with travoprost solution vehicle, 1 drop once daily in the treated eye(s) at night, for 6 weeks
  Interventions: Drug: Dose Level A / Brinzolamide 1% ophthalmic suspension; Drug: Travoprost solution vehicle
- TravB/Brinz (Experimental): Dose Level B / Brinzolamide 1% ophthalmic suspension (fixed combination), 1 drop twice daily in the treated eye(s) morning and night, with travoprost solution vehicle, 1 drop once daily in the treated eye(s) at night, for 6 weeks
  Interventions: Drug: Dose Level B / Brinzolamide 1% ophthalmic suspension; Drug: Travoprost solution vehicle
- TravC/Brinz (Experimental): Dose Level C / Brinzolamide 1% ophthalmic suspension (fixed combination), 1 drop twice daily in the treated eye(s) morning and night, with travoprost solution vehicle, 1 drop once daily in the treated eye(s) at night, for 6 weeks
  Interventions: Drug: Dose Level C / Brinzolamide 1% ophthalmic suspension; Drug: Travoprost solution vehicle
- AZOPT (Active Comparator): Brinzolamide 1% ophthalmic suspension, 1 drop twice daily in the treated eye(s) morning and night, with travoprost solution vehicle, 1 drop once daily in the treated eye(s) at night for 6 weeks
  Interventions: Drug: Brinzolamide 1% ophthalmic suspension AZOPT®; Drug: Travoprost solution vehicle
- TRAV Z (Active Comparator): Brinzolamide suspension vehicle, 1 drop twice daily in the treated eye(s) morning and night, with travoprost 0.004% ophthalmic solution, 1 drop once daily in the treated eye(s) at night, for 6 weeks
  Interventions: Drug: Travoprost 0.004% ophthalmic solution TRAVATAN Z®; Drug: Brinzolamide suspension vehicle
- TRAV Z + AZOPT (Active Comparator): Brinzolamide 1% ophthalmic suspension, 1 drop twice daily in the treated eye(s) twice daily morning and night, with travoprost 0.004% ophthalmic solution, 1 drop once daily in the treated eye(s) at night, for 6 weeks
  Interventions: Drug: Brinzolamide 1% ophthalmic suspension AZOPT®; Drug: Travoprost 0.004% ophthalmic solution TRAVATAN Z®

INTERVENTIONS:
Drug: Dose Level A / Brinzolamide 1% ophthalmic suspension — Fixed combination
  Arms: TravA/Brinz
Drug: Dose Level B / Brinzolamide 1% ophthalmic suspension — Fixed combination
  Arms: TravB/Brinz
Drug: Dose Level C / Brinzolamide 1% ophthalmic suspension — Fixed combination
  Arms: TravC/Brinz
Drug: Brinzolamide 1% ophthalmic suspension AZOPT®
  Other Names: AZOPT®
  Arms: AZOPT; TRAV Z + AZOPT
Drug: Travoprost 0.004% ophthalmic solution TRAVATAN Z®
  Other Names: TRAVATAN Z®
  Arms: TRAV Z; TRAV Z + AZOPT
Drug: Travoprost solution vehicle — Inactive ingredients used for masking purposes
  Arms: AZOPT; TravA/Brinz; TravB/Brinz; TravC/Brinz
Drug: Brinzolamide suspension vehicle — Inactive ingredients used for masking purposes
  Arms: TRAV Z

SUMMARY:
The purpose of this study is to evaluate Travoprost/Brinzolamide fixed combination (Trav/Brinz) administered twice daily as compared to each of its marketed components (TRAVATAN Z® solution and AZOPT® suspension) and to the unfixed combination of TRAVATAN Z® plus AZOPT® in lowering intraocular pressure (IOP).

DETAILED DESCRIPTION:
This study was divided into two phases conducted in sequence. Phase I was the Screening/Eligibility Phase, which included a Screening Visit, followed by two Eligibility Visits. Phase II was the randomized, double-masked, 6-week Treatment Phase which included on-therapy visits at Week 2 and Week 6. Travoprost was administered in 1 of 3 concentration levels (A-C), where A=lowest and C=highest.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with open-angle glaucoma (including open-angle glaucoma with pseudoexfoliation or pigment dispersion) or ocular hypertension;
* IOP within the protocol-specified range at both the Eligibility 1 and 2 Visits. Mean IOP must not be >36 mmHg at any time point;
* Able to understand and sign an informed consent form;
* Other protocol-specified inclusion criteria may apply.

Exclusion Criteria:

* Woman of childbearing potential who is currently pregnant, intends to become pregnant during the study period, breastfeeding, or not using adequate birth control methods to prevent pregnancy throughout the study;
* Unable to discontinue all IOP-lowering ocular medication(s) per the appropriate washout schedule prior to the E1 Visit;
* Chronic, recurrent or severe inflammatory eye disease;
* Ocular trauma within the past 6 months prior to the Screening Visit;
* Ocular infection or ocular inflammation within the past 3 months prior to the Screening Visit;
* Clinically relevant or progressive retinal disease such as retinal degeneration, diabetic retinopathy, or retinal detachment;
* Best-corrected visual acuity (BCVA) score worse than 55 ETDRS letters (equivalent to approximately 0.60 logMAR, 20/80 Snellen, or 0.25 decimal);
* Other ocular pathology (including severe dry eye) that may, in the opinion of the Investigator, preclude the administration of a topical prostaglandin analogue or topical carbonic anhydrase inhibitor;
* Intraocular surgery within the past 6 months prior to the Screening Visit;
* Ocular laser surgery within the past 3 months prior to the Screening Visit;
* Any abnormality preventing reliable applanation tonometry;
* Any other conditions including severe illness which would make the subject, in the opinion of the Investigator, unsuitable for the study;
* History of hepatic or renal disease that would preclude the safe administration of a carbonic anhydrase inhibitor (CAI) in the opinion of the Investigator;
* Hypersensitivity to prostaglandin analogues, topical or oral CAIs, sulfonamide derivatives, or to any component of the study medications in the opinion of the Investigator;
* Recent (within 4 weeks of the Eligibility 1 Visit) use of high dose (> 1 g daily) salicylate therapy;
* Use of any additional topical or systemic ocular hypotensive medication during the study;
* Concurrent use of glucocorticoids administered by any route;
* Less than 30 days stable dosing regimen before the Screening Visit of any medications (excluding the IOP-lowering treatments) or substances administered by any route and used on a chronic basis that may affect IOP (ie, β adrenergic blocking agents);
* Therapy with another investigational agent within 30 days prior to the Screening Visit;
* Other protocol-specified exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 327 (Actual)
Dates: Start 2014-06; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sr. Clinical Manager, GCRA, Pharma, Study Director — Alcon Research

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from 19 study centers located in the US.
Pre-assignment Details: Of the 327 enrolled, 61 subjects were discontinued prior to randomization. This reporting group includes all randomized subjects (266).
Groups:
- TravA/Brinz; TravB/Brinz; TravC/Brinz: Fixed combination, 1 drop twice daily in the treated eye(s) morning and night, with travoprost solution vehicle, 1 drop once daily in the treated eye(s) at night, for 6 weeks
- TRAV Z: Suspension vehicle, 1 drop twice daily in the treated eye(s) morning and night, with travoprost 0.004% ophthalmic solution, 1 drop once daily in the treated eye(s) at night, for 6 weeks
- AZOPT: Ophthalmic suspension, 1 drop twice daily in the treated eye(s) morning and night, with travoprost solution vehicle, 1 drop once daily in the treated eye(s) at night for 6 weeks
- TRAV Z + AZOPT: Ophthalmic suspension, 1 drop twice daily in the treated eye(s) twice daily morning and night, with travoprost 0.004% ophthalmic solution, 1 drop once daily in the treated eye(s) at night, for 6 weeks
Period: Overall Study
Arm/Group | TravA/Brinz | TravB/Brinz | TravC/Brinz | TRAV Z | AZOPT | TRAV Z + AZOPT
Started | 44 | 44 | 44 | 45 | 45 | 44
Completed | 44 | 44 | 44 | 43 | 44 | 43
Not Completed | 0 | 0 | 0 | 2 | 1 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 1 | 1 | 1
Not completed — Lack of Efficacy | 0 | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: This analysis population includes all subjects who were randomized, received study medication, and completed at least 1 scheduled on-therapy study visit.
Groups:
- Total: Total of all reporting groups
Arm/Group | TravA/Brinz | TravB/Brinz | TravC/Brinz | TRAV Z | AZOPT | TRAV Z + AZOPT | Total
Number analyzed (Participants) | 44 | 44 | 44 | 45 | 45 | 43 | 265
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.4 (10.7) | 66.2 (10.4) | 64.4 (11.2) | 64.2 (10.4) | 63.1 (8.4) | 65.3 (10.6) | 64.8 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 26 | 30 | 25 | 23 | 19 | 152
  Male | 15 | 18 | 14 | 20 | 22 | 24 | 113

OUTCOME MEASURES:

1. Primary Outcome: Mean IOP at Week 6
Description: IOP (fluid pressure inside the eye) was assessed using Goldmann applanation tonometry and measured in millimeters of mercury (mmHg). A higher IOP can be a greater risk factor for developing glaucoma or glaucoma progression (leading to optic nerve damage). One eye (study eye) was used for the analysis.
Time Frame: Week 6, 8 AM, 10 AM, 12 PM, 4 PM, and 8 PM
Population: This analysis population includes all subjects who were randomized, received study medication, and completed at least 1 scheduled on-therapy study visit, based upon a last on-therapy carried forward (LOCF) analysis. Here, "n" is the number of subjects with non-missing values at the specific time point for each arm, respectively.
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | TravA/Brinz | TravB/Brinz | TravC/Brinz | TRAV Z | AZOPT | TRAV Z + AZOPT
Number analyzed (Participants) | 44 | 44 | 44 | 45 | 45 | 43
mmHg
  8 AM | 20.2 (0.52) | 18.7 (0.48) | 19.9 (0.58) | 19.3 (0.48) | 22.0 (0.45) | 20.3 (0.72)
  10 AM | 18.9 (0.47) | 17.2 (0.35) | 18.2 (0.55) | 17.4 (0.47) | 19.7 (0.50) | 18.2 (0.59)
  12 PM | 18.9 (0.47) | 17.3 (0.50) | 17.7 (0.51) | 17.2 (0.50) | 19.5 (0.53) | 18.0 (0.57)
  4PM | 18.5 (0.46) | 17.5 (0.43) | 17.3 (0.46) | 17.6 (0.44) | 19.1 (0.50) | 18.0 (0.52)
  8 PM, n=44, 44, 44, 43, 45, 43 | 18.4 (0.43) | 17.5 (0.39) | 17.2 (0.40) | 17.3 (0.43) | 19.3 (0.48) | 18.1 (0.49)

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected for the duration of a subject's participation in the study (up to 11 weeks). AEs were reported as pre-treatment and treatment-emergent.
Description: An AE was defined as any untoward medical occurrence in a subject who was administered a study medication, regardless of whether or not the event had a causal relationship with the medication. AEs were obtained through solicited and spontaneous comments from study subjects, and through observations by the study Investigator.
Groups:
- Pre-treatment: All subjects who signed an informed consent to participate in the study
Arm/Group | TravA/Brinz | TravB/Brinz | TravC/Brinz | TRAV Z | AZOPT | TRAV Z + AZOPT | Pre-treatment
Serious Adverse Events (participants affected / at risk) | 0/44 | 0/44 | 0/44 | 1/45 | 0/45 | 0/44 | 1/327
Other Adverse Events (participants affected / at risk) | 7/44 | 11/44 | 15/44 | 10/45 | 9/45 | 13/44 | 1/327
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TravA/Brinz (N=44) | TravB/Brinz (N=44) | TravC/Brinz (N=44) | TRAV Z (N=45) | AZOPT (N=45) | TRAV Z + AZOPT (N=44) | Pre-treatment (N=327)
Angina unstable (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | TravA/Brinz (N=44) | TravB/Brinz (N=44) | TravC/Brinz (N=44) | TRAV Z (N=45) | AZOPT (N=45) | TRAV Z + AZOPT (N=44) | Pre-treatment (N=327)
Ocular hyperaemia (Eye disorders) | 2 | 8 | 6 | 7 | 0 | 8 | 0
Conjunctival hyperaemia (Eye disorders) | 0 | 3 | 3 | 3 | 3 | 3 | 1
Eye irritation (Eye disorders) | 2 | 2 | 2 | 2 | 3 | 1 | 0
Eye pain (Eye disorders) | 2 | 2 | 3 | 0 | 1 | 1 | 0
Dysgeusia (Nervous system disorders) | 2 | 0 | 3 | 1 | 4 | 3 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.